CLINICAL TRIAL: NCT01318538
Title: Recovery Group for Women With Substance Use Disorders - Stage II Trial
Brief Title: Women's Recovery Group (WRG) Study - A Randomized Controlled Stage II Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Shelly F. Greenfield, Chief Academic Officer; Chief, Division of Women's Mental Health; Kristine M Trustey Endowed Professor of Psychiatry; Director, Clinical and Health Services Research and Education, McLean Hospital; Professor of Psychiatry, Harvard Medical School, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA - 5R01DA015434-05
Record Dates: First submitted 2011-02-22; First posted 2011-03-18 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Substance-Related Disorders; Alcohol-Related Disorders
Keywords: Substance use disorders, Gender differences, women, treatment outcomes, group therapy
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women's Recovery Group (Experimental): The Women's Recovery Group (WRG) is a manual-based group therapy for women heterogeneous with respect to their substance use disorder, co-occurring psychiatric disorders, trauma history, age, and stage of life. The WRG is a 12-session, structured relapse-prevention group therapy that utilizes a cognitive behavioral approach and includes gender-specific content and single-gender group composition. Individual session content was derived from research on gender-specific substance use disorder antecedents, consequences, and treatment outcomes. The overall goals of the treatment are to (1) promote abstinence from all substances including alcohol; (2) improve understanding of specific aspects of SUDs, recovery, and relapse that are relevant to women, and (3) help participants with skills and strategies useful in preventing relapse and promoting recovery.
  Interventions: Behavioral: The Women's Recovery Group
- mixed-gender Group Drug Counseling (Active Comparator): Group Drug Counseling (GDC) is a standard 12-week, 90-minute mixed-gender group therapy. The overall goals of GDC are to 1) help patients to achieve abstinence from all substances including alcohol; 2) educate patients regarding recovery from substance use disorders; 3) increase patients' self-awareness of the problems that their substance use disorder has caused; 4) encourage patients to give mutual support; and 5) help patients learn new ways to cope with problems in order to prevent relapse. The GDC was chosen as the comparison group to approximate group drug counseling that is consistent with treatment as usual within the community.
  Interventions: Behavioral: Group Drug Counseling

INTERVENTIONS:
Behavioral: The Women's Recovery Group — The Women's Recovery Group (WRG) is a manual-based group therapy for women heterogeneous with respect to their substance use disorder, co-occurring psychiatric disorders, trauma history, age, and stage of life. The WRG is a 12-session, structured relapse-prevention group therapy that utilizes a cognitive behavioral approach and includes gender-specific content and single-gender group composition. Individual session content was derived from research on gender-specific substance use disorder antecedents, consequences, and treatment outcomes. The overall goals of the treatment are to (1) promote abstinence from all substances including alcohol; (2) improve understanding of specific aspects of SUDs, recovery, and relapse that are relevant to women, and (3) help participants with skills and strategies useful in preventing relapse and promoting recovery.
  Other Names: WRG
  Arms: Women's Recovery Group
Behavioral: Group Drug Counseling — Group Drug Counseling (GDC) is a standard 12-week, 90-minute mixed-gender group therapy. The overall goals of GDC are to 1) help patients to achieve abstinence from all substances including alcohol; 2) educate patients regarding recovery from substance use disorders; 3) increase patients' self-awareness of the problems that their substance use disorder has caused; 4) encourage patients to give mutual support; and 5) help patients learn new ways to cope with problems in order to prevent relapse. The GDC was chosen as the comparison group to approximate group drug counseling that is consistent with treatment as usual within the community.
  Other Names: GDC
  Arms: mixed-gender Group Drug Counseling

SUMMARY:
The purpose of this Stage II randomized controlled behavioral treatment development trial was to test the effectiveness of the Women's Recovery Group (WRG) relative to mixed-gender Group Drug Counseling (GDC) and demonstrate the feasibility of implementing the WRG in an open-enrollment (i.e., rolling admission) group format at two clinical sites. The Stage II trial aims were to (1) investigate effectiveness of the WRG relative to GDC in a sample of women heterogeneous with respect to substance use and co-occurring psychiatric disorders, and (2) demonstrate the feasibility of implementing WRG in an open enrollment group format characteristic of community treatment programs at two sites.

DETAILED DESCRIPTION:
This Stage II trial builds on the Stage I trial that compared the single-gender WRG to mixed-gender GDC and demonstrated preliminary support for the WRG in treating women with substance use disorders (SUDs). It was hypothesized that women in the WRG would decrease their substance use more so than women in the GDC. The GDC was chosen as the comparison group to approximate group drug counseling that is consistent with treatment as usual within the community. The WRG is a manual-based group therapy for women heterogeneous with respect to their substance dependence, co-occurring psychiatric disorders, trauma history, and age and stage of life. The WRG is a 12-session structured relapse prevention group therapy that utilizes a cognitive-behavioral approach and includes gender-specific content and single-gender group composition. There are 14 specific session topics that can be flexibly implemented in any order for a 12-week sequence of groups. In the Stage I trial, women were randomized to WRG (n=16) or mixed-gender GDC (n =7). No significant differences in outcomes emerged between WRG and GDC during the 12 week group sequence. However, in the 6 months post-treatment, WRG participants showed a pattern of continued reductions in substance use while GDC participants did not. While the design of the Stage I trial was essential for treatment development and testing, the Stage I trial had a small sample size and used a semi-closed enrollment format. However, most treatment is delivered in an open enrollment format (i.e., rolling admission) in which patients enter at any time in the group sequence and exit the group after 12 weeks are completed. Because WRG is intended to be a manual-based treatment ready for dissemination into clinical practice if demonstrated to be effective, the Stage II trial was designed to be implemented in an open group format and to enroll a larger, more diverse sample at two clinical sites. The study was designed to investigate the effectiveness of the WRG relative to the GDC in (1) reducing days of use of any substance from baseline in a sample of women with heterogeneity with regard to their substance dependence, co-occurring psychiatric disorders, and other demographic characteristics, and (2) to demonstrate the feasibility of implementing the WRG in an open-enrollment group format.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were included in the study if they:

  * were 18 years or older
  * used substances within the past 60 days
  * met current Diagnostic and Statistical Manual (DSM)-IV criteria (American Psychiatric Association, 2000; World Health Organization, 1997) of substance dependence (in addition to any nicotine dependence)
  * planned to stay within the area during the study period
  * consented for study personnel to communicate with other mental health professionals from whom they are receiving care
  * furnished the names of two locators who can assist study personnel in locating them during the study period
  * were interested in group treatment
  * lived close enough either to McLean Hospital or SSTAR to come to group weekly
  * were able to sign informed consent.

Exclusion Criteria:

* Patients were excluded if they:

  * had a current medical condition that would prevent regular group attendance
  * had mental retardation or organic mental disorder
  * had certain other major Axis I psychiatric disorders according to the Composite International Diagnostic Interview (CIDI), such as psychotic disorders or bipolar I disorder
  * would be in a residential treatment setting throughout the treatment period in which substance use is monitored and restricted (e.g., a therapeutic community)
  * required medical detoxification (these patients could enter the study after being detoxified)
  * were current intravenous drug users
  * engaged in self-destructive behaviors (e.g., life-threatening bulimia or anorexia, suicide attempts and chronic suicidality) or other behaviors (e.g., violence toward others, assault behaviors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelly F Greenfield, MD, MPH, Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Stanley Street Treatment and Resources (SSTAR), Fall River, Massachusetts

REFERENCES:
- [Background] Greenfield SF, Crisafulli MA, Kaufman JS, Freid CM, Bailey GL, Connery HS, Rapoza M, Rodolico J. Implementing substance abuse group therapy clinical trials in real-world settings: challenges and strategies for participant recruitment and therapist training in the Women's Recovery Group Study. Am J Addict. 2014 May-Jun;23(3):197-204. doi: 10.1111/j.1521-0391.2014.12099.x. PMID 24724875
- [Background] Greenfield SF. Treating Women with Substance Use Disorders: The Women's Recovery Group Manual. New York: Guilford Press; 2016.
- [Result] Greenfield SF, Sugarman DE, Freid CM, Bailey GL, Crisafulli MA, Kaufman JS, Wigderson S, Connery HS, Rodolico J, Morgan-Lopez AA, Fitzmaurice GM. Group therapy for women with substance use disorders: results from the Women's Recovery Group Study. Drug Alcohol Depend. 2014 Sep 1;142:245-53. doi: 10.1016/j.drugalcdep.2014.06.035. Epub 2014 Jul 4. PMID 25042759
- [Result] Sugarman DE, Wigderson SB, Iles BR, Kaufman JS, Fitzmaurice GM, Hilario EY, Robbins MS, Greenfield SF. Measuring affiliation in group therapy for substance use disorders in the Women's Recovery Group study: Does it matter whether the group is all-women or mixed-gender? Am J Addict. 2016 Oct;25(7):573-80. doi: 10.1111/ajad.12443. Epub 2016 Sep 20. PMID 27647710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at McLean Hospital in Belmont, MA and SSTAR Inc. in Fall River, MA using advertisements, flyers, and clinician referrals. At both sites, subjects were recruited from inpatient, residential, partial hospital and outpatient programs. Those recruited from inpatient or residential settings started the groups after discharge.
Pre-assignment Details: Group therapists provided feedback about the groups that they ran, but were not technically enrolled in the study and therefore are not included in initial enrollment number.
Groups:
- Group Therapist: Therapists who ran and led the group sessions for both the single-gender Women's Recovery Group and mixed-gender Group Drug Counseling.
Period: Overall Study
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling | Group Therapist
Started | 52 | 106 | 8
Completed | 52 | 106 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mixed-gender Group Drug Counseling: Group Drug Counseling (GDC) is a standard 12-week, 90-minute mixed-gender group therapy. The overall goals of GDC are to 1) help patients to achieve abstinence from all substances including alcohol; 2) educate patients regarding recovery from substance use disorders; 3) increase patients' self-awareness of the problems that their substance use disorder has caused; 4) encourage patients to give mutual support; and 5) help patients learn new ways to cope with problems in order to prevent relapse. The GDC was chosen as the comparison group to approximate group drug counseling that is consistent with treatment as usual within the community. NOTE: Baseline characteristics reported in Table Below reflect all participants including men assigned to the GDC condition. Analysis of data for study specific aims include only women randomized to WRG (N=52) and GDC (N=48).
- Total: Total of all reporting groups
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling | Total
Number analyzed (Participants) | 52 | 106 | 158
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (12.6) | 47.6 (12.0) | 47 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 0 | 58 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 52 | 105 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 48 | 101 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Marital Status [Number; unit: participants]
  Married | 19 | 41 | 60
  Divorced/Separated | 17 | 27 | 44
  Never married | 12 | 30 | 42
  Unmarried and living with partner | 4 | 5 | 9
  Widowed | 0 | 3 | 3
Education [Number; unit: participants]
  Did not graduate high school | 4 | 7 | 11
  Graduated high school | 7 | 22 | 29
  Some college | 11 | 22 | 33
  Graduated from college | 18 | 34 | 52
  Postgraduate | 12 | 21 | 33
Household Income [Number; unit: participants]
  $0-$20,000 | 17 | 26 | 43
  $20,001-$50,000 | 9 | 31 | 40
  $50,001-$100,000 | 11 | 28 | 39
  More than $100,000 | 15 | 21 | 36
Current psychiatric diagnoses [Number; unit: participants]
  Major depressive disorder | 30 | 58 | 88
  Generalized anxiety disorder | 11 | 20 | 31
  Post-traumatic stress disorder | 9 | 20 | 29
  Any Axis I | 37 | 79 | 116
  Any Axis II | 9 | 15 | 24
Substance use diagnoses [Number; unit: participants]
  Alcohol current | 43 | 97 | 140
  Alcohol lifetime | 45 | 101 | 146
  Cocaine current | 8 | 20 | 28
  Cocaine lifetime | 17 | 40 | 57
  Cannabis current | 3 | 16 | 19
  Cannabis lifetime | 7 | 27 | 34
  Opioids current | 7 | 19 | 26
  Opioids lifetime | 13 | 27 | 40
  Sedatives current | 5 | 11 | 16
  Sedatives lifetime | 5 | 17 | 22
Substance use days (past 30 days) [Mean (Standard Deviation); unit: Days]
  Alcohol use days | 12.7 (9.9) | 15.4 (10.5) | 14.6 (10.3)
  Days of any substance use (including alcohol) | 16.5 (9.3) | 17.8 (9.8) | 17.3 (9.6)
  Drug use days (excluding alcohol) | 4.8 (9.2) | 4.8 (9.0) | 4.8 (9.0)
  Primary substance use days | 13.4 (9.9) | 15.7 (10.4) | 14.9 (10.3)
  Heavy drinking days | 9.8 (9.7) | 13.5 (10.6) | 12.3 (10.6)
  Drinks per drinking day | 7.0 (5.0) | 11.3 (7.1) | 10.0 (6.8)
  Controlled environment days | 0.38 (1.6) | 0.26 (1.3) | .30 (1.4)
Addiction Severity Index (ASI) composite scores [Mean (Standard Deviation); unit: units on a scale from 0-1] — The Addiction Severity Index (ASI) is a multidimensional assessment of substance-related problems which yields composite scores for alcohol use, drug use, psychiatric status, medical status, legal status, family/social relationships, and employment status. Composite scores range from 0 to 1, with higher scores indicating more significant problems.
  units on a scale from 0-1
    Alcohol | 0.47 (0.33) | 0.55 (0.29) | 0.52 (0.30)
    Drug | 0.07 (0.11) | 0.08 (0.15) | 0.08 (0.13)
    Medical | 0.18 (0.24) | 0.18 (0.27) | 0.18 (0.26)
    Psychiatric | 0.25 (0.20) | 0.19 (0.19) | 0.21 (0.19)
    Legal | 0.04 (0.11) | 0.09 (0.68) | 0.07 (0.56)
    Family | 0.29 (0.55) | 0.24 (0.28) | 0.26 (0.39)
    Employment | 0.42 (0.24) | 0.43 (0.29) | 0.43 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Mean Days of Any Substance Use for Women
Description: This represents the percent change from baseline in the mean number of days per month of any substance use (i.e. drug and/or alcohol) for women. Days of substance use was assessed using the Timeline Follow-Back at baseline and then monthly for 9 months. The In-Treatment phase includes months 1-3, the 3 Month Post-Treatment phase includes months 4-6, and the 6 Month Post-Treatment phase includes months 7-9. The in-treatment and 2 post-treatment phases were compared to baseline data of mean days of any substance use. Outcomes were analyzed using loglinear (negative binomial) regression models with estimation via generalized estimating equations (GEE). The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction.
Time Frame: In-treatment (months 1-3), 3 Month Post-treatment (months 4-6), 6 Month Post-Treatment (months 7-9)
Population: Only women were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: % change in mean substance use days
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
% change in mean substance use days
  In-treatment Phase (months 1-3) | -76.5 [-83.9 to -65.7] | -76.5 [-85.0 to -63.0]
  3 Month Post-treatment Phase (months 4-6) | -68.4 [-76.9 to -56.8] | -73.3 [-83.0 to -58.1]
  6 Month Post-Treatment Phase (months 7-9) | -62.2 [-74.9 to -41.3] | -70.8 [-80.5 to -56.1]
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction.The study was powered for the primary analysis concerning treatment group differences in the degree of improvement in the number of days of any substance use and in the Addiction Severity Index (ASI) composite scores. With a total of 100 women, the study was adequately powered to detect a minimum 5 day benefit in the # of days of any substance use (power = 83%); Test type: Superiority or Other; p = 0.821, loglinear (negative binomial) regression; Analyzed using loglinear (negative binomial) regression models with estimation via generalized estimating equations (relative changes i.e. % change)

2. Secondary Outcome: Percent Change in Mean Alcohol Use Days for Women
Description: This represents the percent change from baseline in the mean number of alcohol use days. Days of alcohol use was assessed using the Timeline Follow-Back at baseline and then monthly for 9 months. The In-Treatment phase includes months 1-3, the 3 Month Post-Treatment phase includes months 4-6, and the 6 Month Post-Treatment phase includes months 7-9. The in-treatment and 2 post-treatment phases were compared to baseline alcohol use data. Outcomes were analyzed using loglinear (negative binomial) regression models with estimation via generalized estimating equations (GEE). The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction.
Time Frame: In-treatment (months 1-3), 3 Month Post-treatment (months 4-6), 6 Month Post-Treatment (months 7-9)
Population: Some participants did not complete this measure at the specified time points. Only women were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: percent change in Alcohol Use Days
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
percent change in Alcohol Use Days
  In-treatment Phase (months 1-3) | -80.6 [-87.5 to -69.9] | -82.6 [-89.7 to -67.2]
  3 Month Post-treatment Phase (months 4-6) | -70.3 [-79.1 to -57.6] | -80.5 [-88.6 to -66.6]
  6 Month Post-Treatment Phase (months 7-9) | -67.8 [-80.5 to -46.8] | -80.4 [-87.7 to -68.5]
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction. Note: Women in both WRG and GDC groups had significant (p<0.0001 reductions in mean # of alcohol use days during treatment (9.9 and 12.4 day reductions for WRG and GDC respectively) and at 6 months post-treatment (8.3 and 12.2 day reductions); Test type: Superiority or Other; p = 0.519, loglinear (negative binomial) regression; We used loglinear (negative binomial) regression models with estimation via generalized estimating equations (GEE)

3. Primary Outcome: Change in Mean ASI Alcohol Composite Score for Women
Description: This represents the change from baseline in mean ASI Alcohol composite scores. The ASI was administered at baseline, at months 1-6, and then at month 9. The In-Treatment phase includes months 1-3, the 3 Month Post-Treatment phase includes months 4-6, and the 6 Month Post-Treatment phase includes months 7-9. The in-treatment and 2 post-treatment phases were compared to baseline ASI data. Outcomes were analyzed using linear mixed effect models. These models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction.
  The ASI is a multidimensional assessment of substance-related problems which yields composite scores for alcohol use, drug use, psychiatric status, medical status, legal status, family/social relationships, and employment status. Composite scores range from 0 to 1, with higher scores indicating more significant problems.
Time Frame: In-treatment (months 1-3), 3 Month Post-treatment (months 4-6), 6 Month Post-Treatment (months 7-9)
Population: Only women were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: change in ASI Alcohol composite score
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
change in ASI Alcohol composite score
  In-treatment Phase (months 1-3) | -0.27 [-0.33 to -0.22] | -0.33 [-0.39 to -0.28]
  3 Month Post-treatment Phase (months 4-6) | -0.28 [-0.34 to -0.22] | -0.36 [-0.43 to -0.30]
  6 Month Post-Treatment Phase (months 7-9) | -0.30 [-0.39 to -0.21] | -0.35 [-0.44 to -0.26]
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction. The study was powered for the primary analysis concerning treatment group differences in the degree of improvement in the number of days of any substance use and in the Addiction Severity Index (ASI) composite scores.With 100 women (50 in each treatment group), the study was adequately powered to detect a 0.2 benefit in the ASI drug and alcohol composite scores (power = 94%); Test type: Superiority or Other; p = 0.253, Linear mixed effect models; This measure was analyzed using using linear mixed effect models with estimation via restricted maximum likelihood (absolute changes in the mean)

4. Primary Outcome: Change in Mean ASI Drug Composite Score for Women
Description: This represents the change from baseline in mean ASI Drug composite scores. The ASI was administered at baseline, at months 1-6, and then at month 9. The In-Treatment phase includes months 1-3, the 3 Month Post-Treatment phase includes months 4-6, and the 6 Month Post-Treatment phase includes months 7-9. The in-treatment and 2 post-treatment phases were compared to baseline ASI data. Outcomes were analyzed using linear mixed effect models. These models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction.
  The ASI is a multidimensional assessment of substance-related problems which yields composite scores for alcohol use, drug use, psychiatric status, medical status, legal status, family/social relationships, and employment status. Composite scores range from 0 to 1, with higher scores indicating more significant problems.
Time Frame: In-treatment (months 1-3), 3 Month Post-treatment (months 4-6), 6 Month Post-Treatment (months 7-9)
Population: Only women were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: change in ASI Drug composite score
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
change in ASI Drug composite score
  In-treatment Phase (months 1-3) | -0.03 [-0.05 to -0.02] | -0.03 [-0.05 to -0.01]
  3 Month Post-treatment Phase (months 4-6) | -0.03 [-0.05 to -0.01] | -0.03 [-0.05 to -0.01]
  6 Month Post-Treatment Phase (months 7-9) | -0.02 [-0.05 to 0.02] | -0.04 [-0.07 to 0.00]
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.667, Linear mixed effect models; [statistical method as in outcome 3, analysis 1]

5. Other Pre Specified Outcome: Therapist Adherence
Description: All therapists were female to eliminate any therapist-patient gender matching effects. There were eight therapists in total: 4 who led WRG groups and 4 who led GDC groups. All group sessions were videotaped each week so that we could measure therapist adherence to the treatment they were assigned to. Two independent raters completed adherence scales for a random selection of 20% of WRG and 10%of GDC sessions. For both groups, the extensiveness to which the therapist engaged in a behavior during the session was rated with a 5-point Likert scale (0 = not at all; 4 = extensively). Adherence scores were calculated by averaging all scores for each question (25 questions for WRG; 18 for GDC) on the measure. The scores reported here represent the average of all WRG therapists scores from all session, and all GDC therapist scores from all sessions. Scores range from 0 to 4.
Time Frame: In treatment (weeks 1-12)
Measure: Mean (Standard Deviation); unit: units on a 0-4 adherence scale
Units Other Than Participants: Sessions
Groups:
- Women's Recovery Group: Participants in this analysis are the therapists that lead the WRG groups. The Women's Recovery Group (WRG) is a manual-based group therapy for women heterogeneous with respect to their substance use disorder, co-occurring psychiatric disorders, trauma history, age, and stage of life. The WRG is a 12-session, structured relapse-prevention group therapy that utilizes a cognitive behavioral approach and includes gender-specific content and single-gender group composition. Individual session content was derived from research on gender-specific substance use disorder antecedents, consequences, and treatment outcomes. The overall goals of the treatment are to (1) promote abstinence from all substances including alcohol; (2) improve understanding of specific aspects of SUDs, recovery, and relapse that are relevant to women, and (3) help participants with skills and strategies useful in preventing relapse and promoting recovery.
- Mixed-gender Group Drug Counseling: Participants in this analysis are the therapists that lead GDC groups. Group Drug Counseling (GDC) is a standard 12-week, 90-minute mixed-gender group therapy. The overall goals of GDC are to 1) help patients to achieve abstinence from all substances including alcohol; 2) educate patients regarding recovery from substance use disorders; 3) increase patients' self-awareness of the problems that their substance use disorder has caused; 4) encourage patients to give mutual support; and 5) help patients learn new ways to cope with problems in order to prevent relapse. The GDC was chosen as the comparison group to approximate group drug counseling that is consistent with treatment as usual within the community.
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 4 | 4
Number analyzed (Sessions) | 28 | 27
units on a 0-4 adherence scale | 3.8 (0.13) | 3.6 (0.28)

6. Other Pre Specified Outcome: Group Attendance
Description: Treatment attendance was calculated by summing the number of treatment sessions attended. Therefore, numbers range from 0-12.
Time Frame: In treatment (weeks 1-12)
Population: Only women were included in this analysis.
Measure: Mean (Standard Deviation); unit: sessions attended
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
sessions attended | 7.64 (1.36) | 7.69 (1.36)
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

7. Other Pre Specified Outcome: Group Stability
Description: Treatment group stability was calculated using the Percentage of Group Change Index which captures change in group membership composition from session to session separately for each individual within each group (specific to the calendar period that each person was in the group). The value can range from 0 (i.e., the exact same membership from one session to the next) to 1 (i.e., complete turnover in membership). The average values across all sessions were taken to get an overall sense of the amount of turnover each person experienced in the group during the period in calendar time they were in treatment.
Time Frame: In treatment (weeks 1-12)
Population: Only women were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
units on a scale | 0.39 (0.07) | 0.36 (0.07)
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

8. Secondary Outcome: Percent Change in Mean Drug Use Days for Women
Description: This represents the percent change from baseline in the mean number of drug use days (excluding alcohol) for women. Days of drug use was assessed using the Timeline Follow-Back at baseline and then monthly for 9 months. The In-Treatment phase includes months 1-3, the 3 Month Post-Treatment phase includes months 4-6, and the 6 Month Post-Treatment phase includes months 7-9. The in-treatment and 2 post-treatment phases were compared to baseline data of mean drug use days. Outcomes were analyzed using loglinear (negative binomial) regression models with estimation via generalized estimating equations (GEE). The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction.
Time Frame: In-treatment (months 1-3), 3 Month Post-treatment (months 4-6), 6 Month Post-Treatment (months 7-9)
Population: Only women were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: % change in mean drug use days
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
% change in mean drug use days
  In-treatment Phase (months 1-3) | -66.3 [-85.5 to -21.8] | -40.8 [-62.4 to -6.8]
  3 Month Post-treatment Phase (months 4-6) | -76.7 [-89.6 to -47.5] | -51.1 [-71.9 to 16.3]
  6 Month Post-Treatment Phase (months 7-9) | -62.2 [-83.0 to -15.9] | -41.9 [-71.7 to 19.2]
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction. Note: Women in both WRG and GDC groups had significant (p<0.05) reductions in mean number of drug use days during treatment (3.0 and 1.5 day reductions for WRG and GDC respectively); however at 6 months post-treatment, the reductions were significant for WRG (2.8 day reduction; p<0.05) but not for GDC (1.5 day reduction; p>0.01); Test type: Superiority or Other; p = 0.464, loglinear (negative binomial) regression; We used loglinear (negative binomial) regression models with estimation via generalized estimating equations (GEE)

9. Secondary Outcome: Percent Change in Mean Heavy Drinking Days for Women
Description: This represents the percent change from baseline in the mean number of heavy drinking days for women. Number of heavy drinking days was assessed using the Timeline Follow-Back at baseline and then monthly for 9 months. The In-Treatment phase includes months 1-3, the 3 Month Post-Treatment phase includes months 4-6, and the 6 Month Post-Treatment phase includes months 7-9. The in-treatment and 2 post-treatment phases were compared to baseline data of mean heavy drinking days. Outcomes were analyzed using loglinear (negative binomial) regression models with estimation via generalized estimating equations (GEE). The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction.
Time Frame: In-treatment (months 1-3), 3 Month Post-treatment (months 4-6), 6 Month Post-Treatment (months 7-9)
Population: Only women were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: % change in mean heavy drinking days
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
% change in mean heavy drinking days
  In-treatment Phase (months 1-3) | -89.6 [-91.4 to -81.8] | -85.7 [-92.7 to -72.0]
  3 Month Post-treatment Phase (months 4-6) | -82.4 [-89.5 to -70.4] | -82.0 [-90.0 to -67.5]
  6 Month Post-Treatment Phase (months 7-9) | -83.8 [-91.2 to -70.3] | -83.2 [-90.2 to -71.2]
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction. Note: Women in both WRG and GDC groups had significant (p<0.0001) reductions in mean number of heavy drinking days during treatment (8.6 and 12.1 days reduction for WRG and GDC, respectively) and at 6 months post-treatment (8.0 and 11.8 day reductions); Test type: Superiority or Other; p = 0.904, loglinear (negative binomial) regression; We used loglinear (negative binomial) regression models with estimation via generalized estimating equations (GEE)

10. Secondary Outcome: Change in Mean Drinks Per Drinking Day for Women
Description: This represents the change from baseline in the mean number of drinks per drinking day. Drinks per drinking day was assessed using the Timeline Follow-Back at baseline and then monthly for 9 months. The In-Treatment phase includes months 1-3, the 3 Month Post-Treatment phase includes months 4-6, and the 6 Month Post-Treatment phase includes months 7-9. The in-treatment and 2 post-treatment phases were compared to baseline data of mean drinks per drinking day. Outcomes were analyzed using loglinear (negative binomial) regression models with estimation via generalized estimating equations (GEE). The models included the effects of treatment group, phase (3 levels), and the treatment group by phase interaction.
Time Frame: In-treatment (months 1-3), 3 Month Post-treatment (months 4-6), 6 Month Post-Treatment (months 7-9)
Population: Only women were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: change in mean drinks per drinking day
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 52 | 48
change in mean drinks per drinking day
  In-treatment Phase (months 1-3) | -1.96 [-3.77 to -0.16] | -2.87 [-4.74 to -1.01]
  3 Month Post-treatment Phase (months 4-6) | -1.47 [-3.91 to 0.98] | -1.41 [-3.99 to 1.18]
  6 Month Post-treatment Phase (months 7-9) | -1.22 [-4.57 to 2.13] | -0.76 [-4.28 to 2.76]
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; The models included the effects of treatment group, phase (3 levels), and the treatment by phase interaction. Note: Women in both the WRG and GDC groups had significant (p<0.05) reductions in mean number of drinks per drinking day only during the in treatment phase (2.0 and 2.9 reductions for WRG and GDC, respectively); Test type: Superiority or Other; p = 0.799, linear mixed effect model; [statistical method as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over a period of 1 year and 9 months (November 2009 to August 2011).
Description: Adverse events were collected between November of 2009 and August 2011, during which participants were either in treatment or completing 3-month and 6-month post-treatment assessments.
Groups:
- Women's Recovery Group: The WRG is a manual-based group therapy for women heterogeneous with respect to their substance dependence, co-occurring psychiatric disorders, trauma history, and age and stage of life. The WRG is a 12-session, structured relapse-prevention group therapy that utilizes a cognitive behavioral approach and includes gender-specific content and single-gender group composition. Individual session content was derived from research on gender-specific substance use disorder antecedents, consequences, and treatment outcomes. The overall goals of the treatment are to (1) promote abstinence from all substances including alcohol; (b) improve understanding of specific aspects of SUDs, recovery, and relapse that are relevant to women, and (c) help participants with skills and strategies useful in preventing relapse and promote recovery.
- Mixed-gender Group Drug Counseling: The GDC is a standard 12-week, 90-minute mixed-gender group therapy. The overall goals of GDC are to 1) help patients to achieve abstinence from all substances including alcohol; 2) educate patients regarding recovery from substance dependence; 3) increase patients' self-awareness of the problems that substance dependence has caused; 4) encourage patients to give mutual support; and 5) help patients learn new ways to cope with problems in order to prevent relapse.
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Serious Adverse Events (participants affected / at risk) | 4/52 | 13/106
Other Adverse Events (participants affected / at risk) | 13/52 | 8/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women's Recovery Group (N=52) | Mixed-gender Group Drug Counseling (N=106)
Dehydration (General disorders) | 0 | 1 — Participant hospitalized for dehydration; unrelated to study
Seizure (Nervous system disorders) | 0 | 1 — Participant had a seizure and went to the emergency department; unrelated to study
Overdose (General disorders) | 0 | 2 — One participant overdosed on Lyrica and required a visit to the emergency department; another participant overdosed on heroin and was admitted to the hospital for one night. Both were unrelated to the study
Colon Surgery (Surgical and medical procedures) | 1 | 0 — Participant was hospitalized for colon surgery; unrelated to study
Hospitalization (Gastrointestinal disorders) | 1 | 1 — One participant was hospitalized for an intestinal obstruction; another participant was hospitalized for bleeding ulcers. Both were unrelated to the study
Chest Pain (General disorders) | 1 | 0 — Participant experienced chest pain and was admitted to the hospital for observation; unrelated to study
Abscess (Skin and subcutaneous tissue disorders) | 1 | 0 — Participant had abscess on leg; unrelated to study
Post-Surgery Infection (Infections and infestations) | 0 | 1 — Participant had surgery and was hospitalized overnight for a post-surgery infection; unrelated to study
Stroke (Nervous system disorders) | 0 | 1 (2) — Participant had a stroke twice; unrelated to study
Heart Attack (Cardiac disorders) | 0 | 1 — Participant was hospitalized for a heart attack; unrelated to study
Death - Heart Attack (Cardiac disorders) | 0 | 2 — Two participants passed away from a heart attack; both were unrelated to the study
Death - Stroke (Nervous system disorders) | 0 | 1 — Participant passed away from a stroke; unrelated to study
Hospitalization (General disorders) | 0 | 1 — Participant was hospitalized for anemia; unrelated to study
Back Pain (Nervous system disorders) | 0 | 1 — Participant hurt his back, went to the emergency department, and was admitted to the hospital. He was later diagnosed with sciatica; unrelated to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Women's Recovery Group (N=52) | Mixed-gender Group Drug Counseling (N=106)
Acute Asthma Episode (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — One participant required a hospital visit; the other required an overnight hospitalization
Alcohol Intoxication (General disorders) | 0 | 1 — Required a visit to the emergency department
Gastrointestinal Virus Hospitalization (Gastrointestinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Required a visit to the emergency department
Fainting Episode (General disorders) | 0 | 1 — Required a hospitalization
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Required a visit to the emergency department
Surgical Procedure - Removal of Lymph Nodes (Surgical and medical procedures) | 1 | 0
Ovarian Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Required a hospitalization
Motor Vehicle Accident (Social circumstances) | 1 | 0 — Required a hospitalization
Hospitalization (General disorders) | 1 | 0 — Participant was hospitalized for risk of suicide
Gastrointestinal Discomfort (Gastrointestinal disorders) | 2 | 0 — Required a visit to the emergency department
Broken Arm (Musculoskeletal and connective tissue disorders) | 1 | 1 — Required a visit to the emergency department
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 — Required a visit to the emergency department
Animal Bite (Infections and infestations) | 1 | 0 — Participant received IV antibiotics for cat bite in the emergency department
Involuntary Psychiatric Hospitalization (Psychiatric disorders) | 1 | 0
Dehydration (General disorders) | 0 | 1 — Required a visit to the emergency department

LIMITATIONS AND CAVEATS:
* relatively small sample
* sample was almost all white and well-educated (questionable generalizability)
* therapists not blind to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No